CLINICAL TRIAL: NCT01712308
Title: A Phase-2, Prospective, Open-Label Study to Determine the Safety and Efficacy of Sotatercept (ACE-011) in Subjects With Myeloproliferative Neoplasm (MPN) -Associated Myelofibrosis and Anemia
Brief Title: Sotatercept in Treating Patients With Myeloproliferative Neoplasm-Associated Myelofibrosis or Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0534; NCI-2012-03139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0534 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-10-18; First posted 2012-10-23 (Estimated); Results first posted 2023-06-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Anemia; Myelodysplastic/Myeloproliferative Neoplasm; Myelofibrosis
MeSH Terms: conditions — Anemia; Myelodysplastic-Myeloproliferative Diseases; Primary Myelofibrosis | interventions — ACE-011; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Monotherapy (sotatercept) (Experimental): Patients receive sotatercept SC once every 3 weeks. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients unable to achieve anemia-response after 8 cycles will be taken off study.
  Interventions: Biological: Sotatercept
- Treatment combination (Ruxolitinib + sotatercept) (Experimental): patients that are already on therapy with ruxolitinib (for at least for 6 months, and on stable dose for last 2 months) will continue ruxolitinib in addition to sotatercept SC once every 3 weeks. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients unable to achieve anemia-response after 8 cycles will be taken off study.
  Interventions: Biological: Sotatercept; Drug: Ruxolitinib

INTERVENTIONS:
Biological: Sotatercept — Given SC
  Other Names: ACE-011; Decoy Activin Receptor ACE-011
Drug: Ruxolitinib
  Other Names: INCB018424
  Arms: Treatment combination (Ruxolitinib + sotatercept)

SUMMARY:
This phase II trial studies the side effects of and how well sotatercept works in treating patients with myeloproliferative neoplasm-associated myelofibrosis or anemia. Sotatercept may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
The goal of this clinical research study is to learn if sotatercept can help to control MPN-associated myelofibrosis and anemia. The safety of this drug will also be studied.

OUTLINE: This is a dose-escalation study.

Patients receive sotatercept subcutaneously (SC) once every 3 weeks. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients unable to achieve anemia-response after 8 cycles will be taken off study.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* MPN-associated myelofibrosis
* Anemic patient OR red blood cell (RBC)-transfusion-dependent patient
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) and aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) equal to or less than 2.5 x upper limit of normal (ULN), or equal to or less than 4 x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to myelofibrosis [MF])
* Direct bilirubin equal to or less than 1.5 x ULN; or equal to or less than 2 x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis related to MF)
* Creatinine clearance equal to or more than 50 mL/min
* Treatment-related toxicities from prior therapies must have resolved to grade equal to or less than 1
* Women of childbearing potential and men must agree to using medically approved (i.e., mechanical or pharmacological) contraceptive measure for at least 112 days following the last dose of sotatercept (ACE-011); males must agree to use a latex condom or non-latex condom NOT made of natural (animal) membrane during any sexual contact with females of childbearing potential or a pregnant female while participating in the study and for at least 112 days following the last dose of sotatercept (ACE-011), even if he has a vasectomy
* For cohort of patients that are already on ruxolitinib therapy: on therapy with ruxolitinib for at least for 6 months, and on stable dose for last 2 months, before starting therapy with sotatercept

Exclusion Criteria:

* Serious medical condition or psychiatric illness that would prevent, (as judged by the treating physician) the subject from signing the informed consent form or any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or lactating female
* Known positive for human immunodeficiency virus-1 (HIV-1), or active infection with hepatitis-B or -C
* Use of any MPN-associated myelofibrosis-directed therapy within 2 weeks prior to study day 1 (other than ruxolitinib at a stable dose for patients in the combination cohort as stated in inclusion criteria)
* Symptomatic congestive heart failure, unstable angina, or unstable cardiac arrhythmia
* Prior sotatercept
* Major surgery within 4 weeks prior to day 1
* Severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product
* Uncontrolled hypertension (systolic blood pressure [SBP] equal to or more than 140 or diastolic blood pressure [DBP] equal to or more than 90)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prithviraj Bose, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Combination (Ruxolitinib + Sotatercept): patients that are already on therapy with ruxolitinib (for at least for 6 months, and on stable dose for last 2 months) will continue ruxolitinib in addition to sotatercept SC once every 3 weeks. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients unable to achieve anemia-response after 8 cycles will be taken off study.
  Sotatercept: Given SC
  Ruxolitinib
Period: Overall Study
Arm/Group | Treatment Monotherapy (Sotatercept) | Treatment Combination (Ruxolitinib + Sotatercept)
Started | 35 | 21
Completed | 35 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Monotherapy (Sotatercept) | Treatment Combination (Ruxolitinib + Sotatercept) | Total
Number analyzed (Participants) | 35 | 21 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 4 | 18
  >=65 years | 21 | 17 | 38
Age, Continuous [Median (Full Range); unit: years] | 66 [47 to 83] | 71 [47 to 84] | 67 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 21 | 14 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 29 | 14 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 35 | 21 | 56

OUTCOME MEASURES:

1. Primary Outcome: Anemia-response
Description: Defined as an increase in hemoglobin level equal to or greater than 1.5 g/L without red blood cell-transfusion OR becoming red blood cell-transfusion-independent in a patient who is red blood cell-transfusion-dependent. Will be based on the intent-to-treat principle.
Time Frame: Up to 84 days
Population: Of the 35 participants on the monotherapy arm, 27 were evaluable for response. Of the 21 participants on the Combination Therapy arm, 19 were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Monotherapy (Sotatercept) | Treatment Combination (Ruxolitinib + Sotatercept)
Number analyzed (Participants) | 27 | 19
Participants | 8 | 6

2. Primary Outcome: Duration of Response
Description: Response date to loss of response or last follow up.
Time Frame: Up to 9 years
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment Monotherapy (Sotatercept) | Treatment Combination (Ruxolitinib + Sotatercept)
Number analyzed (Participants) | 27 | 19
Months | 23.3 [3.9 to 68.4] | 19.9 [3.7 to 56.8]

ADVERSE EVENTS:
Time Frame: Up to 9 years
Arm/Group | Treatment Monotherapy (Sotatercept) | Treatment Combination (Ruxolitinib + Sotatercept)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/21
Serious Adverse Events (participants affected / at risk) | 11/35 | 10/21
Other Adverse Events (participants affected / at risk) | 30/35 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Monotherapy (Sotatercept) (N=35) | Treatment Combination (Ruxolitinib + Sotatercept) (N=21)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Chest wall pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 2 (3)
Lung infection (Infections and infestations) | 0 (0) | 3 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Non cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain in extremity (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Monotherapy (Sotatercept) (N=35) | Treatment Combination (Ruxolitinib + Sotatercept) (N=21)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Cardiac disorders (Cardiac disorders) | 5 (7) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 8 (8)
Dizziness (Nervous system disorders) | 6 (8) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3
Edema limbs (General disorders) | 9 (9) | 3 (3)
Elevated Albumin/Creatinine Ratio (Investigations) | 4 (4) | 1 (1)
elevated transaminase levels (Investigations) | 1 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Fatigue (General disorders) | 6 (6) | 3 (3)
Fever (General disorders) | 3 (3) | 3 (5)
Flu like symptoms (General disorders) | 9 (28) | 14 (31)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 10 (17) | 9 (14)
Headache (General disorders) | 2 (3) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (7) | 5 (5)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (7) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (5) | 1 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (5)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 9 (16) | 6 (11)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 16 (34) | 9 (22)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral neuropathy (Nervous system disorders) | 4 (4) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 10 (13) | 7 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 8 (9) | 5 (10)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5) | 1 (1)
Weight loss (Investigations) | 2 (2) | 1 (1)
Bleeding Hemorrhage (General disorders) | 8 (13) | 6 (10)
Psychiatric Disorders (Psychiatric disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT01712308/Prot_SAP_000.pdf